CLINICAL TRIAL: NCT03617770
Title: A Sleep Intervention to Improve Glycemic Control and Reduce Diabetes Distress in Working Adults With Type 1 Diabetes
Brief Title: A Sleep Intervention in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Chicago (Other)
Responsible Party: Principal Investigator, Pamela Martyn-Nemeth, Assistant Professor Biobehavioral Health Science College of Nursing, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0762; P30DK092949 (NIH)
Record Dates: First submitted 2018-07-13; First posted 2018-08-06 (Actual); Results first posted 2021-03-05 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Short Sleep Phenotype; Type1diabetes
Keywords: type 1 diabetes; glycemic control; sleep; diabetes distress
MeSH Terms: conditions — Sleep Wake Disorders; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Sleep optimization intervention will be compared to a healthy living attention control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep-Opt-In (Experimental): Sleep optimization intervention
  Interventions: Behavioral: Sleep Opt-In
- Healthy Living (Active Comparator): Health education
  Interventions: Behavioral: Healthy Living

INTERVENTIONS:
Behavioral: Sleep Opt-In — 8-week intervention that includes a wearable sleep tracker, didactic content, smartphone application and counseling
  Arms: Sleep-Opt-In
Behavioral: Healthy Living — 8-week intervention that includes weekly telephone counseling on healthy living.
  Arms: Healthy Living

SUMMARY:
Insufficient sleep and sleep irregularity (variability in sleep duration) are increasingly recognized as important contributors to glucose control and diabetes distress in type 1 diabetes (T1D). Up to 40% of adults with T1D had a sleep duration less than 6-6.5 hours per night. Diabetes distress is reported (40% prevalence) in individuals with T1D and is associated with poor glucose control. Despite findings that sleep disturbances are common in T1D, the current understanding of the effects of strategies to improve sleep on diabetes distress, and glucose control is limited. The purpose of this pilot study is to evaluate the effects of a sleep intervention on sleep duration, diabetes distress and glucose control in individuals with T1D and habitual short sleep. A randomized controlled trial in 20 adults aged 18 to 65 years with T1D is proposed. Eligible participants will be randomly assigned to a sleep intervention group or a control group. Differences between the two groups on the outcomes of sleep duration, diabetes distress and glucose control will be evaluated. Findings from this proposed pilot study will serve as the foundation for a larger clinical trial to improve sleep, reduce diabetes distress, and improve glucose control.

DETAILED DESCRIPTION:
Insufficient sleep and sleep irregularity (variability in sleep duration) are increasingly recognized as important contributors to glycemic control and diabetes distress in type 1 diabetes (T1D). Up to 40% of adults with T1D had a sleep duration < 6-6.5 hours per night, either by self-report or objectively assessed actigraphy. Diabetes distress is reported (40% prevalence) in individuals with T1D and is associated with poor glycemic control. Despite findings that sleep disturbances are common in T1D, the current understanding of the effects of sleep optimization on sleep, diabetes distress, and glycemic control is limited. The purpose of this pilot and feasibility trial is to evaluate the effects of a T1D-specific sleep optimization intervention (Sleep-Opt-In) on the outcomes of sleep, diabetes distress and glycemic control in individuals with T1D and habitual short sleep. The specific aims are to determine if Sleep-Opt-In will: 1) be feasible and acceptable to the target population; 2) result in improved sleep duration and regularity; 3) result in improved glycemic control; and 4) lower diabetes distress. To achieve these aims, a randomized controlled trial in 20 adults aged 18 to 65 years with T1D is proposed. Participants will be screened for habitual sleep duration < 6.5 hours per night. Eligible subjects will be randomized to the T1D-Sleep-Opt-In group or attention control group. A one-week run-in period is planned, with baseline measures of sleep (duration and regularity), glycemia (A1C, fructosamine, glycemic variability), and diabetes distress (Diabetes Distress Scale). The T1D-Sleep-Opt-In will entail a novel technology-assisted behavioral sleep extension intervention developed to leverage rapidly increasing public interest in sleep tracking by consumers (+500% in 3 years). This technology employs four elements: a wearable sleep tracker, didactic content, an interactive smartphone application, and brief telephone counseling. The intervention will be T1D-specific by addressing T1D-related sleep issues such as nocturnal hypoglycemia. The attention control group will participate in a healthy living information program. At completion (Week 8) and post-program (Weeks 12 and 24), baseline measures will be repeated to determine differences between the two groups and sustainability of the intervention. Findings from this proposed pilot study will serve as the foundation for a larger clinical trial to improve sleep, reduce diabetes distress, and improve glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes for one year or more
* self-reported habitual sleep duration less than 6.5 hours per night during work- or weekdays
* own a smartphone.

Exclusion Criteria:

* insomnia
* sleep apnea
* severe hypoglycemia within past 6 months
* treated with an insulin pump with hybrid closed-loop features
* rotating shift or night shift work
* estimated glomerular filtration rate less than 45 ml/min
* heart failure
* cirrhosis
* chronic obstructive pulmonary disease requiring oxygen
* actively treated for cancer or psychiatric problem
* history of stroke
* pregnant or planning pregnancy
* HbA1c 10% or higher.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Martyn-Nemeth, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sleep-Opt-In | Healthy Living
Started | 9 (9) | 5 (5)
Completed | 8 (8) | 5
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sleep-Opt-In | Healthy Living | Total
Number analyzed (Participants) | 9 | 5 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 5 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.1 (7.1) | 30.0 (7.6) | 30.1 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 8 | 3 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Sleep Duration
Description: change in minutes of sleep (actigraphy-derived)
Time Frame: Assessing change between two time points:Week 0 to week 8
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sleep-Opt-In | Healthy Living
Number analyzed (Participants) | 5 | 3
minutes | 385 (40) | 388 (39)

2. Primary Outcome: Sleep Regularity
Description: Change in sleep regularity (variability)
Time Frame: Assessing change between two time points: from week 0 to week 8
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sleep-Opt-In | Healthy Living
Number analyzed (Participants) | 5 | 3
minutes | 46 (20) | 56 (8)

3. Secondary Outcome: HbA1c
Description: HbA1c (A1C%)
Time Frame: Change between two time points, week 0 to week 8
Measure: Mean (Standard Deviation); unit: % of glucose saturation on hemoglobin
Arm/Group | Sleep-Opt-In | Healthy Living
Number analyzed (Participants) | 5 | 3
% of glucose saturation on hemoglobin | 6.48 (0.74) | 6.7 (1.4)

4. Secondary Outcome: Glucose Variability
Description: Change in glucose variability (CV%) (continuous glucose monitor derived)
Time Frame: Assessing change between two time points: from week 0 to week 8
Measure: Mean (Standard Deviation); unit: percentage of CV
Arm/Group | Sleep-Opt-In | Healthy Living
Number analyzed (Participants) | 5 | 3
percentage of CV | 34.4 (4.6) | 31.6 (5.0)

5. Secondary Outcome: Diabetes Distress
Description: Change in Diabetes Distress Scale score, 6-point, 17-item Likert scale. The 17 items are summed. The sum score is divided by 17 to provide a mean item score. Higher scores indicate greater distress. Score interpretation:
  < 2.0 = little distress 2.0-2.9 = moderate distress 3.0 or greater = hah distress
Time Frame: Assessing change between two time points: from week 0 to week 8
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Sleep-Opt-In | Healthy Living
Number analyzed (Participants) | 5 | 3
change in score on a scale | 1.2 (0.23) | 3.1 (1.36)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Sleep-Opt-In | Healthy Living
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/5
Other Adverse Events (participants affected / at risk) | 0/9 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT03617770/Prot_SAP_000.pdf